CLINICAL TRIAL: NCT01979588
Title: How Does the Clinical Tool 'What's Going Around' Affect Clinical Practice
Acronym: WGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Ari Robiscek, Vice President for Clinical and Quality Informatics, Associate CMIO, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: What's Going Around
Record Dates: First submitted 2013-10-30; First posted 2013-11-08 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Influenza Like Illness; Asthma; Group A Streptococcal Infection; Pertussis
MeSH Terms: conditions — Asthma; Streptococcal Infections; Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Providers do not have access to What's Going Around Tool but receive an instructional video explaining tool
  Interventions: Other: Control
- What's Going Around Tool (Active Comparator): Provider has access to What's Going Around Tool. Provider also shown a video explaining how to use Tool
  Interventions: Other: What's Going Around tool

INTERVENTIONS:
Other: What's Going Around tool — Provider has access to the What's Going Around tool
  Arms: What's Going Around Tool
Other: Control — Provider does not have access to the What's Going Around tool but received information regarding the tool prior to study initiation
  Arms: Control

SUMMARY:
Previous work has shown that the epidemiological context of a patient's presentation can provide important information for clinicians to aid in diagnosis and treatment. With current electronic health records, it is increasingly possible to perform syndromic surveillance that is local and specific to a patient's characteristics.

The investigators have developed algorithms for syndromic surveillance for a number of conditions in which contextual information might be of use to treating clinicians. The syndromic surveillance algorithms already developed are for influenza-like-illness, whooping cough, asthma exacerbation, Group A Streptococcal pharyngitis, and gastroenteritis infection.

The investigators plan on studying these tools with a clustered randomized control cohort study evaluating how clinical decision making is affected by use of these tools by outpatient general practitioners. The goal is to incorporate these validated algorithms into a quality improvement tool which will provide point-of-care clinical decision support to clinicians

DETAILED DESCRIPTION:
The epidemiological context of a patient's presentation can provide important information for clinicians to aid in diagnosis and treatment. The investigators previously developed and validated a syndromic surveillance tool for detecting influenza-like illness (ILI) encounters. The investigators then evaluated 40,642 outpatient ILI episodes during 'flu seasons' over 6 years. The investigators found that even after controlling for patient presentation and physician factors, the context in which a patient presented was strongly associated with the likelihood that an antimicrobial agent would be prescribed. Specifically, patients were less likely to be prescribed an antibiotic if they presented with ILI during the pandemic influenza period (when awareness of 'flu season' was very high), or after their physician had personally seen many patients with ILI in the prior week.

Currently, most clinicians have only limited access to data regarding the 'context' in which a patient presents. Under such circumstances, physicians are often unaware of local epidemiological information that could help them make optimal treatment decisions. In centers with advanced use of electronic health records (EHRs), it is increasingly possible to perform syndromic surveillance that is local (e.g. specific to a neighborhood or school district), current (e.g. updated daily), and specific to a patient's characteristics (e.g. age, chief complaint).

To that end, the investigators have developed algorithms for syndromic surveillance for a number of syndromes including Asthma, ILI, Pertussis, Group A Streptococcus Pharyngitis, and Gastroenteritis. These algorithms may provide contextual information that might be of use to clinicians.

The purpose of this study is to determine the effect of how a point-of-care clinical decision tool in the form of syndromic surveillance algorithms affect clinical decision making amongst outpatient health care providers and also patient outcomes. We will be using a 2 year look back prior to tool roll out as a comparison.

Specific Aims:

To determine the effect this point-of-care clinical decision tool has on clinical decision making amongst primary care providers.

To determine the clinical outcomes of patients whose physicians had access to these tools

To understand how these point-of-care clinical decision tools are used among healthcare providers in day to day practice

ELIGIBILITY:
Inclusion Criteria:

All patients seen in a Northshore University HealthSystem outpatient clinic (Family Medicine, Internal Medicine or Pediatric) between the Nov 1 2013 to Oct 31 2014

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 206703 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of visits for ILI in which a patient was prescribed an antibacterial agent during the seasonal flu season | 1 year

SECONDARY OUTCOMES:
Percentage of visits for ILI in which a patient was prescribed an antiviral agent during the seasonal flu season | 1 year
Percent of primary care visits in which a patient received an antibiotic | 1 year

OTHER OUTCOMES:
Percentage of visits for pediatric patients with asthma in which asthma counseling performed | 1 year
Percent of time a pertussis PCR was sent for patients with a complaint of cough during a period of high pertussis prevalence | 1 year
Percent of pharyngitis patients who received a Group A Strep test during a period of high prevalence of group A strep | 1 year
Percent of time that a pertussis active antibiotic was prescribed in a patient with a complaint of a cough during a period of high pertussis prevalence | 1 year
Percent of pharyngitis patients who received a Group A Strep test during a period of low prevalence of group A strep | 1 year
Percent of pharyngitis patients who received a Group A strep appropriate antibiotic during a period of high prevalence of group A strep | 1 year
Percent of pharyngitis patients who received a Group A Strep appropriate antibiotic during a period of low prevalence of group A strep | 1 year
Percent of patients with asthma who have a hospital visit for asthma | 1 year
Percentage of days that a physician used the What's Going Around tool of all days he/she worked in a year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ari Robicsek, MD, Principal Investigator — Endeavor Health
Locations (1):
- Northshore University HealthSystem, Evanston, Illinois, United States

REFERENCES:
- [Background] Hebert C, Beaumont J, Schwartz G, Robicsek A. The influence of context on antimicrobial prescribing for febrile respiratory illness: a cohort study. Ann Intern Med. 2012 Aug 7;157(3):160-9. doi: 10.7326/0003-4819-157-3-201208070-00005. PMID 22868833